CLINICAL TRIAL: NCT06116032
Title: Immune Profiling for Cancer Immunotherapy Response
Status: Recruiting | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Brock C. Christensen, Professor of Epidemiology, Molecular and Systems Biology, and of Community and Family Medicine, Dartmouth-Hitchcock Medical Center
Other Study IDs: Study02001227
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Tumor, Solid; Hematologic Malignancy; Blood Cancer
Keywords: Immunotherapy
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and FFPE tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Standard of Care Checkpoint: Patients receiving standard of care FDA approved immunotherapy
  Interventions: Diagnostic Test: Methylation Cytometry
- Bone Marrow Transplant: Patients undergoing transplant for hematologic malignancy
  Interventions: Diagnostic Test: Methylation Cytometry
- CAR T: Patients undergoing CAR T therapy
  Interventions: Diagnostic Test: Methylation Cytometry

INTERVENTIONS:
Diagnostic Test: Methylation Cytometry — Assessment of the ability of Methylation Cytometry in pre-treatment peripheral blood and in repeated measures over the duration of treatment to predict treatment response or occurrence of adverse events.

SUMMARY:
In patients clinically treated with FDA-approved immunotherapy the investigators will assess the predictive value of pre- and on-treatment 1) immune-methylation profiling across cancer types, and 2) immune-methylation profiling and cytokine profiling within cancer types.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients receiving or will receive immunotherapy under FDA- approved indication (e.g. checkpoint inhibitor therapy with pembrolizumab, nivolumab, or ipilimumab, or cellular immunotherapy).
* Participants are eligible regardless of the type of prior therapy (i.e. prior immunotherapy treated participants can be included).

Exclusion Criteria:

* Pregnant women/fetuses/neonates
* Prisoners
* Decision-impaired individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients who will receive or who are receiving immunotherapy under FDA- approved indication
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Response to therapy | 5 years
  The investigators will employ iRECIST, and outcome criteria will be clinically evaluated and include the primary endpoints of progression (non-responders) or response, with patients followed up every month for 6 months (or until death, loss to follow-up, or withdrawal of consent), judged according to the objective response rate (ORR) assessed using iRECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Brock C Christensen, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided